CLINICAL TRIAL: NCT06872892
Title: A Phase III, Randomised, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of BI 1291583 2.5 mg Administered Once Daily for up to 76 Weeks in Patients With Bronchiectasis (The AIRTIVITY™ Study)
Brief Title: The AIRTIVITY™ Study: A Study to Find Out Whether BI 1291583 Helps People With Bronchiectasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397-0014; 2024-518589-29-00 (Registry Identifier: EU CTIS); U1111-1317-2315 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental)
  Interventions: Drug: BI 1291583
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib
  Arms: Treatment arm
Drug: Placebo matching BI 1291583 — Placebo matching BI 1291583
  Arms: Placebo arm

SUMMARY:
This study is open to adults and adolescents aged 12 to under 18 with bronchiectasis. People can participate in this study if they produce sputum and have had flare-ups (also called exacerbations).

The purpose of this study is to find out whether a medicine called BI 1291583 helps people with bronchiectasis. Participants are put into 2 groups randomly, which means by chance. One group takes BI 1291583 tablets and the other group takes placebo tablets. A placebo tablet looks like the BI 1291583 tablet but does not contain any medicine. Participants take 1 tablet once a day for up to 1 year and 6 months.

Participants are in the study for up to 1 year and 8 months. During this time, participants visit the study site up to 10 times and get about 13 phone calls from the site staff. Participants regularly complete a diary on a smartphone about their bronchiectasis symptoms and study doctors regularly check for any changes. The study doctors document when participants experience flare-ups. The number of flare-ups is compared between the participants who receive BI 1291583 and those who receive the placebo. The study doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

* Male or female participants. Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per International Council of Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1 % per year when used consistently and correctly, as well as one barrier method. A list of contraception methods meeting these criteria is provided in the participant information.
* Signed and dated written informed consent and assent, if applicable, prior to admission to the study, in accordance with GCP and local legislation.
* Age of participants when signing the informed consent/assent ≥12 years.

  -- Adolescents need to weigh at least 35 kg at Visit 1.
* Clinical history consistent with bronchiectasis (e.g. cough, chronic sputum production, recurrent respiratory infections) and investigator confirmed diagnosis of bronchiectasis by CT scan where bronchiectasis has been documented by a radiologist.

Participants whose past CT scan image records are not available will undergo a chest CT scan during Screening. Historical scans must not be older than five years.

* Adult participants should be able to produce sputum for Pseudomonas aeruginosa assessment during the screening period.
* History of documented pulmonary exacerbations requiring antibiotic treatment. In the 12 months before Visit 1, participants must have had either:

  * at least 2 exacerbations, or
  * at least 1 exacerbation and an St. George's Respiratory Questionnaire (SGRQ) Symptoms score of >40 at screening Visit 1 (adults only)
  * at least 1 exacerbation and high symptom burden according to the investigator's judgement (adolescents only) For participants on oral or inhaled antibiotics as chronic treatment for bronchiectasis and participants on Cystic Fibrosis Transmembrane Conductance Regulator Modulator Therapy (CFTR-MT), at least one exacerbation must have occurred since initiation of antibiotics or CFTR-MT.

Exclusion criteria:

* Any new or newly diagnosed condition of primary or secondary immunodeficiency within 1 year before randomisation.
* Allergic bronchopulmonary aspergillosis being treated or requiring treatment.
* Tuberculosis or non-tuberculosis mycobacterial infection being treated or requiring treatment
* Any findings in the medical examination and/or laboratory value assessed at Screening Visit 1 or during screening period, that in the opinion of the investigator may put the participant at risk by participating in the trial.
* Any clinically relevant (at the discretion of the investigator) acute respiratory infection or ongoing pulmonary exacerbation at screening visit or during the screening unless recovered in the opinion of the investigator prior to Visit 2.
* Any relevant pulmonary, gastrointestinal, hepatic, renal, cardiovascular, metabolic, immunological, hormonal, or other disorder that, in the opinion of the investigator, may put the participant at risk by participating in the study.
* Major surgery (major according to the investigator's assessment) performed within 6 weeks prior to randomisation or scheduled during trial period.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated in situ non-melanoma skin cancers or in situ carcinoma of uterine cervix.
* Evidence or medical history of moderate or severe liver disease (Child-Pugh score B or C hepatic impairment).
* estimated Glomerular Filtration Rate (eGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (adults) or Chronic Kidney Disease Under 25 (CKiD-U25) (adolescents) <30 mL/min at Visit 1.
* Previous treatment with a dipeptidyl peptidase-1 (DPP1) (Cathepsin C (CatC)) inhibitor. (Note: Participants that were randomised and only received placebo in studies with DPP1 (CatC) inhibitor are allowed.) Further exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1755 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-09-14 (Estimated); Study Completion 2028-10-12 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of adjudicated pulmonary exacerbations (number of events per person year) up to Week 76 | up to 76 weeks

SECONDARY OUTCOMES:
Time to first adjudicated pulmonary exacerbation up to Week 76 | up to 76 weeks
Absolute change from baseline in Quality of Life Questionnaire - Bronchiectasis (QOL-B) respiratory symptoms domain score at Week 52 (participants ≥ 16 years) | at baseline, at week 52
  The QOL-B is a patient reported outcome (PRO) measure assessing symptoms, functioning and health-related quality of life of patients with bronchiectasis. It consists of 37 items covering the following domains: respiratory symptoms, physical functioning, vitality, role functioning, health perception, emotional functioning, social functioning, and treatment burden.
  All items are rated on a 4-point response scale ranging from 'a lot' to 'not at all' with the recall period 'the previous week'. Domain scores are generated ranging from 0 to 100, with higher scores indicating less symptom burden, better functioning, and higher health-related quality of life respectively.
Absolute change from baseline in post-bronchodilator Forced Expiratory Volume in the first second (FEV1) %pred at Week 52 | at baseline, at week 52
Absolute change from baseline in post-bronchodilator Forced Vital Capacity (FVC) %pred at Week 52 | at baseline, at week 52
Annualised rate of severe adjudicated pulmonary exacerbations up to Week 76 | up to 76 weeks
Time to first adjudicated severe pulmonary exacerbation up to Week 76 | up to 76 weeks

CONTACTS AND LOCATIONS:
Locations (496):
- United States (79):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Medical Group Alaska, Anchorage, Alaska
  - Dignity Health, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Newport Native MD, Inc, Newport Beach, California
  - Paradigm Clinical Research - Redding, Redding, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Ventura County Medical Center, Ventura, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, North Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - Meris Clinical Research-Brandon-69466, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Essence MD Research, Naples, Florida
  - Premier Medical Associates, The Villages, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland St. Joseph Medical Group Pulmonary Care and Sleep Medicine, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Health Partners Specialty, Saint Paul, Minnesota
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Medical College - Hawthorne, Hawthorne, New York
  - Northwell Health, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Stern Research Partners, LLC, Huntersville, North Carolina
  - Pinehurst Medical Clinic, Inc. - East, Pinehurst, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - ProMedica Physicians Pulmonary and Sleep Medicine - Toledo, Toledo, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Health Honickman Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Horizon Clinical Research Group, Cypress, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Metroplex Pulmonary & Sleep Center, McKinney, Texas
  - Methodist Heart and Lung Institute, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Element Research Group, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Vermont, Burlington, Vermont
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Virginia Commonwealth University Health Systems, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (12):
  - Centro Dr. Lazaro Langer S.R.L, Alberdi Sur
  - CEC- Centro de Especialidades Cardiovasculares, Bahía Blanca
  - Hospital Aleman, CABA
  - Centro de Investigación Clinica Belgrano, CABA
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Mautalen- Salud e Investigacion, CABA
  - Equipo Ciencia, CABA
  - APRILLUS-Asistencia e Investigacion, Ciudad Autonoma Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata
  - Centro Respiratorio de Quilmes, Quilmes
  - Instituto de Especialidades de la Salud Rosario, Rosario
  - Ibamedica, Santa Fe
- Australia (16):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Heart of Australia Research Institute, Chelmer, Queensland
  - Lung Research Queensland, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Peninsula Health, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Trialswest, Spearwood, Western Australia
- Austria (4):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Hospital Hietzing, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Vitaz - Campus Sint-Niklaas, Sint-Niklaas
- Brazil (8):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Chronos Pesquisa Clinica, Brasília
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - Mecas Servicos Educacionais e Administrativos LTDA, João Pessoa
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Netspiro Clinica Medica Ltda - Respsono, São Bernardo do Campo
  - INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo
- Bulgaria (9):
  - MHAT Rahila Angelova AD, Pernik
  - Medical Center Unimed, Plovdiv
  - SHATPPD "Dr. Dimitar Gramatikov", Rousse
  - Multiprofile Hospital MHATEM 'Pirogov', Sofia, Sofia
  - Diagnostics And Consultation Center Convex Ltd., Sofia
  - Medical Center "Pulmovision", Sofia
  - Medical Center Tara, Veliko Tarnovo
  - Medical Center "Sveti Ivan Rilski", Vidin
  - Sbalpfz-Vratsa, Vratsa
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - Cardio 1 Medical Clinic, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - BLC Clinical Research, Burlington, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Diex Recherche (Sherbrooke Est), Sherbrooke, Quebec
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
  - Royal University Hospital (Saskatoon), Saskatoon, Saskatchewan
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Chile (2):
  - Centro de Estudios Clínicos CEC, Santiago
  - Centro de Investigación del Maule, Talca
- China (51):
  - China-Japan Friendship Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guizhou People's Hospital, Guiyang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huzhou Central Hospital, Huzhou
  - Jiangmen Central Hospital, Jiangmen
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanjing First Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - The Children's Hospital of Fudan University, Shanghai
  - Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou People's Hospital, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Wuxi People's Hospital, Wuxi
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yixing People'S Hospital, Yixing
- Croatia (3):
  - Specialty Hospital Medico, Rijeka
  - Clinical Hospital Centar Sestre Milosrdnice, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - MediTrial s.r.o., Jindřichův Hradec
  - University Hospital Motol, Prague
  - The First Pulmonary Private Practice, Prague
- Denmark (5):
  - Aalborg Sygehus Syd, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Hvidovre Hospital, Hvidovre
  - Copenhagen University Hospital, Rigshospitalet, København Ø
  - Vejle University Hospital, Vejle
- Egypt (4):
  - CRC-Alexandria University, Alexandria
  - Ain Shams University Clinical Research Center (MASRI), Cairo
  - Air Force Specialized Hospital, Cairo
  - Kasr Al Aini, Cairo University, Cairo
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital / TYKS, Turku
- France (11):
  - CHU Amiens-Picardie, Amiens
  - HOP Intercommunal, Créteil
  - INS Coeur Poumon, Lille
  - Hopital De La Croix-Rousse, Lyon
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - Hôpital Cochin, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Pontchaillou, Rennes
  - HOP Nord Laennec, Saint-Herblain
  - Hôpital Larrey - CHU de Toulouse, Tououse
- Germany (32):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Velocity Clinical Research Germany GmbH, Ahrensburg, Ahrensburg
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Universitätsklinikum Bonn AöR, Bonn
  - Augustiner Krankenhäuser GmbH, Cologne
  - Universitätsklinikum Köln (AöR), Cologne
  - Caritas-Krankenhaus St. Maria gGmbH, Donaustauf
  - Klinikum Dortmund gGmbH, Dortmund
  - Technische Universität Dresden, Dresden
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München AÖR, München
  - Pneumologisches Studienzentrum München-West, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Westbrandenburg GmbH, Potsdam
  - Helios Hanseklinikum Stralsund, Stralstund
  - BAG Wiesbaden, Wiesbaden
- Hong Kong (2):
  - Prince of Wales Hospital-Hong Kong-20715, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (3):
  - Koranyi National Institute For Pulmonolgy, Budapest
  - BKS Research Ltd, Hatvan
  - Da Vinci Private Clinic, Pécs
- India (8):
  - Jawahar Lal Nehru Medical College, Ajmer
  - M. S. Ramaiah Institute of Health Science, Bengaluru
  - Narayana Health - Mazumdar Shaw Medical Center, Bengaluru
  - B. P. Poddar Hospital and Medical Research Limited, Kolkata
  - Midland Healthcare & Research Center, Lucknow
  - Siddhi Hospital, C/o Dr. Mutha Hospital, Nashik
  - Pandit Bhagwat Dayal Sharma Post Graduate Institute of Medical Sciences, Rohtak
  - Government Hospital for Chest and Communicable Diseases (GHCCD), Visakhapatnam
- Ireland (3):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - Connolly Hospital Blanchardstown, Dublin
- Israel (4):
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (17):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Policlinico S. Orsola-Malpighi, Bologna
  - AOU Policlinico G. Rodolico San Marco, Catania
  - Azienda Ospedaliera San Martino, Genova
  - Istituto G. Gaslini, Genova
  - A.O.U.Policlinico G.Martino, Messina
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Di Monza, Monza (MB)
  - A.O. dei Colli, Napoli
  - AOU San Luigi Gonzaga, Orbassano (TO)
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Policlinico "Paolo Giaccone", Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Osp. Pediatrico Bambin Gesù, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (38):
  - Nagoya University Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - Chiba University Hospital, Chiba, Chiba
  - Kameda Clinic, Chiba, Kamogawa
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Fukuoka Children's Hospital, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Terada Clinic, Respiratory Medicine & General practice, Hyogo, Himeji
  - University of Tsukuba Hospital, Ibaraki, Tsukuba
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Minami Kyoto Hospital, Kyoto, Joyo
  - Kyoto University Hospital, Kyoto, Kyoto
  - Matsusaka City Hospital, Mie, Matsusaka
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Oita University Hospital, Oita, Yufu
  - Kurashiki Central Hospital, Okayama, Kurashiki
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Toneyama Medical Center, Osaka, Toyonaka
  - Saga University Hospital, Saga, Saga
  - Saitama Cardiovascular and Respiratory Center, Saitama, Kumagaya
  - Shiga University of Medical Science Hospital, Shiga, Otsu
  - Matsue Medical Center, Shimane, Matsue
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Tenryu Hospital, Shizuoka, Hamamatsu
  - Tokushima University Hospital, Tokushima, Tokushima
  - Institute of Science Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Fukujuji Hospital, Tokyo, Kiyose
  - Toranomon Hospital, Tokyo, Minato-ku
  - National Center for Child Health and Development, Tokyo, Setagaya-ku
  - Keio University Hospital, Tokyo, Shinjuku-ku
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
  - Yamaguchi University Hospital, Yamaguchi, Ube
- Kazakhstan (2):
  - Multidisciplinary City Hospital №1 of the Akimat of Astana, Astana
  - Regional Clinical Hospital of the Health Department of the Karaganda Region, Karaganda
- Latvia (7):
  - Med.Center OLVI Health Center Assotiation,Private Practice, Daugavpils
  - Daugavpils Regional Hospital LTD Centre Outpatient Clinic, Daugavpils
  - VCA Dubultu Medical center, Jūrmala
  - Riga 1st Hospital, Riga
  - LUMPII Doctors practice, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East University Hospital, Upeslejas
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Republic Klaipeda Hospital, Klaipėda
  - Vilnius University Hospital, Santariskiu, Vilnius
  - Inmedica, Vilnius
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Setar, Kedah
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Hospital Raja Perempuan Zainab II, Kelantan
  - Institut Perubatan Respiratori, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Mexico (10):
  - Centro de Investigacion Integral MEDIVEST S.C, Chihuahua City
  - Mediadvance Clinical S.A.P.I de C.V., Chihuahua City
  - Centro de Investigacion Farmacologica del Bajío, S.C., León
  - Soluciones terapeuticas medico quirurgicas S de RL de CV, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - Oaxaca Site Management Organization, S.C., Oaxaca City
  - Asociación Mexicana para la Investigacion Clínica, A.C(AMIC), Pachuca
  - Clinical Research Institute S.C., Tlalnepantla
  - Arke SMO S.A. de C.V., Veracruz de Ignacio de La Llave
- Netherlands (6):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
  - Haga Ziekenhuis, The Hague
  - UMC Utrecht, Utrecht
  - Gelre Ziekenhuis Zutphen, Zutphen
- New Zealand (7):
  - NZ Respiratory and Sleep Institute, Greenlane East, Auckland
  - Momentum clinical Research Tauranga, Tauranga, Bay of Plenty
  - Momentum Clinical Research Dunedin, Dunedin, Otago
  - Waikato Hospital, Hamilton, Waikato Region
  - Momentum Clinical Research, Mount Cook, Wellington Region
  - Christchurch Hospital, Christchurch
  - Middlemore Clinical Trials, Papatoetoe
- Philippines (5):
  - Iloilo Doctors Hospital, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Health Cube Medical Clinics, Mandaluyong
  - Quirino Memorial Medical Center, Quezon City
  - Philippine General Hospital, Taft, Manila
- Poland (6):
  - Respiratory Medicine Centre, private prac., Bialystok, Bialystok
  - M2M Med Sp. z o.o. sp. j., Chorzów
  - Screenmed Sp. z o.o., Piaseczno
  - EMED, Center of Medical Services,Private Prac,Rzeszow, Rzeszów
  - Altamed Specjalistyczna Praktyka Lekarska Pawel Sliwinski, Warsaw
  - Medical Center K2J2, Wołomin
- Portugal (7):
  - ULS da Região de Aveiro, Aveiro
  - ULS Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS do Alto Ave, Guimarães
  - ULS da Região de Leiria, E.P.E., Leiria
  - ULS de Santa Maria, E.P.E, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
- Puerto Rico (3):
  - San Juan Bautista School of Medicine, Caguas
  - VA Caribbean Healthcare System, San Juan
  - Puerto Rico Consortium for Clinical Investigation, San Juan
- Romania (4):
  - Marius Nasta Institute of Pneumophthisiology, Bucharest
  - SC Medlife S.A, Cluj-Napoca
  - Clinical Hospital of Pneumophysiology Leon Daniello, Cluj-Napoca
  - Clinical Hospital Of Infectious Diseases And Pneumophysiology Dr.Victor Babes Timisoara, Timișoara
- Singapore (4):
  - National University Hospital-Singapore-42005, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (2):
  - Univ. Hospital Martin, Martin
  - Plucna ambulancia Hrebenar s.r.o., Spišská Nová Ves
- South Africa (5):
  - Iatros International, Bloemfontein
  - Dr Ismail Abdullah, Cape Town
  - Addington Hospital, Durban
  - Enhancing Care Foundation NPC, Mount Edgecombe
  - CAPRISA Offices on the King DinuZulu Hospital Complex, Springfield
- South Korea (18):
  - Hallym University Sacred Heart Hospital, Anyang
  - Chungbuk National University Hospital, Chungju
  - Yeongnam University Hospital, Daegu
  - Ulsan University Hospital, Dong-gu Ulsan
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Jeonbuk National University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (21):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Infanta Elena, Huelva
  - Hospital Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital de Mérida, Mérida
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Puerto Real, Puerto Real
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sweden (3):
  - Universitetssjukhuset, Örebro, Örebro
  - Karolinska University Hospital, Stockholm
  - CTC Clinical Trial Consultants AB, Uppsala
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - University Hospital of Lausanne, Lausanne
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
  - National Taiwan University Hospital Yun-Lin Branch, Yunlin County
- Thailand (5):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Songklanagarind Hospital, Songkhla
  - King Chulalongkorn Memorial Hospital, Thailand
- Turkey (Türkiye) (8):
  - Sağlık Bilimleri Üniversitesi Gülhane Eğitim ve Araştırma Hastanesi, Ankara
  - Ankara University Medical Faculty, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Adnan Menderes Üniversitesi, Aydin
  - Istanbul University Medical Faculty Capa Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Manisa Celal Bayar Üniversitesi Tıp Fakültesi, Manisa
  - Mersin University Research and Training Hospital Chest Diseases Department, Yenişehir
- United Kingdom (23):
  - Belfast City Hospital, Belfast
  - Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Bradford Royal Infirmary, Bradford
  - Velocity Clinical Research, Bristol, Bristol
  - Royal Papworth Hospital, Cambridge
  - University Hospital Llandough, Cardiff
  - Ninewells Hospital & Medical School, Dundee, Scotland
  - University Hospital Hairmyres, East Kilbride
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Hospital for Children and Young People, Edinburgh
  - Western General Hospital, Edinburgh
  - Freeman Hospital, High Heaton
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Liverpool Heart & Chest Hospital, Liverpool
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - Craigavon Area Hospital, Portadown
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com